CLINICAL TRIAL: NCT00311363
Title: A Long-Term Study of XP13512 Versus Placebo Treatment Assessing Maintenance of Efficacy and Safety in Patients With Restless Legs Syndrome.
Brief Title: Long-Term Study of Gabapentin Enacarbil (GEn, XP13512) vs. Placebo in Patients With Restless Legs Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111461; XP060 (Other: XenoPort, Inc.)
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Results first posted 2011-05-25 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2011-05

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — 1-(((alpha-isobutanoyloxyethoxy)carbonyl)aminomethyl)-1-cyclohexaneacetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GEn (XP13512) 1200 mg (Experimental): GEn (XP13512) 1200 mg
  Interventions: Drug: GEn (XP13512)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GEn (XP13512) — 1200 mg GEn (XP13512) orally, once daily for 24 weeks followed by either 1200 mg GEn (XP13512) or placebo, orally, once daily for an additional 12 weeks
  Other Names: Gabapentin Enacabil; XP13512
  Arms: GEn (XP13512) 1200 mg
Drug: GEn (XP13512) — 1200 mg GEn (XP13512), orally, once daily for 24 weeks followed by either 1200 mg GEn (XP13512) or placebo, orally, once daily for an additional 12 weeks
  Other Names: Gabapentin Enacarbil; XP13512
  Arms: GEn (XP13512) 1200 mg
Drug: Placebo — Placebo, orally, once daily for 12 weeks following single blind 24-week phase
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to assess the maintenance of efficacy of gabapentin enacarbil (GEn, XP13512) taken once daily in the long-term treatment of patients suffering from Restless Legs Syndrome (RLS).

DETAILED DESCRIPTION:
This study was a multicenter, blinded, randomized withdrawal study in subjects with primary Restless Legs Syndrome (RLS). Eligible subjects were initially enrolled in a 24-week single blind (SB) treatment period during which they received XP13512. Subjects who completed the initial treatment period and met the responder criteria were then randomized 1:1 to receive either XP13512 or placebo during the 12-week double-blind (DB) treatment period. The primary study objective was to assess the maintenance of efficacy of XP13512 1200 mg taken once daily in the long-term treatment of subjects with primary RLS. The secondary study objectives were to assess maintenance of improvements in sleep outcomes and quality of life, and to assess the safety and tolerability of XP13512 in the treatment of primary RLS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary RLS, based on the International RLS Study Group Diagnostic Criteria.

Exclusion Criteria:

* A sleep disorder (e.g., sleep apnea) that may significantly affect the assessment of RLS;
* Neurologic disease or movement disorder (e.g., diabetic neuropathy, Parkinson's disease, Multiple Sclerosis, dyskinesias, and dystonias);
* Abnormal laboratory results, electrocardiogram (ECG) or physical findings;
* Pregnant or lactating women;
* Women of childbearing potential who are not practicing an acceptable method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2006-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] Bogan RK, Bornemann MA, Kushida CA, Tran PV, Barrett RW; XP060 Study Group. Long-term maintenance treatment of restless legs syndrome with gabapentin enacarbil: a randomized controlled study. Mayo Clin Proc. 2010 Jun;85(6):512-21. doi: 10.4065/mcp.2009.0700. PMID 20511481

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 27 participants who completed the Single-blind Treatment Period who either elected not to enroll into the Double-blind Treatment Period or were considered non-responders and were not randomized.
Groups:
- Single-blind (SB) GEn 1200 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262) 1200 milligrams (mg) once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 168: two ER tablets (total dose of 1200 mg GEn).
- DB Placebo: Days 169 to 182: one 600 mg ER tablet of GEn and one matching placebo tablet for a 2-week blinded taper period. Days 183 to 252: two blinded placebo tablets. Days 253 to 260, participants tapered to one placebo tablet.
- DB GEn 1200 mg: Days 169 to 252: two 600 mg ER tablets (1200 mg GEn). Days 253 to 260, participants tapered to one 600 mg ER tablet.
Period: 24-Week Single-Blind Treatment Period
Arm/Group | Single-blind (SB) GEn 1200 mg | DB Placebo | DB GEn 1200 mg
Started | 327 | 0 | 0
Completed | 221 | 0 | 0
Not Completed | 106 | 0 | 0
Not completed — Adverse Event | 42 | 0 | 0
Not completed — Lack of Efficacy | 13 | 0 | 0
Not completed — Withdrawal by Subject | 27 | 0 | 0
Not completed — Lost to Follow-up | 12 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0
Not completed — Elective Surgery | 1 | 0 | 0
Not completed — Work Shift Changed to Evenings | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Period: 12-Week Double-Blind Treatment Period
Arm/Group | Single-blind (SB) GEn 1200 mg | DB Placebo | DB GEn 1200 mg
Started | 0 | 98 | 96
Completed | 0 | 84 | 84
Not Completed | 0 | 14 | 12
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 6 | 4
Not completed — Withdrawal by Subject | 0 | 2 | 4
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Per Sponsor, Unknown | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Single-blind (SB) Safety Population: subjects who received at least 1 dose of SB study drug
  1 subject withdrew from the SB period prior to receiving drug due to protocol non-compliance, and thus was excluded from the SB-Safety Population
Groups:
- SB GEn 1200 mg: Oral gabapentin enacarbil (GEn; XP13512/GSK1838262) 1200 milligrams (mg) once daily. Days 1 to 3: one extended release (ER) tablet (600 mg GEn). Days 4 to 168: two ER tablets (total dose of 1200 mg GEn).
- Total: Total of all reporting groups
Arm/Group | SB GEn 1200 mg | DB Placebo | DB GEn 1200 mg | Total
Number analyzed (Participants) | 326 | 98 | 96 | 520
Age Continuous [Mean (Standard Deviation); unit: Years] — The Safety Population (all participants who received at least one dose [or any portion of a dose] of study drug) was used for all baseline characteristics.
  Years | 49.8 (12.38) | 52.2 (12.07) | 50.7 (11.68) | 51.5 (11.87)
Sex: Female, Male [Count of Participants; unit: Participants] — The Safety Population (all participants who received at least one dose [or any portion of a dose] of study drug) was used for all baseline characteristics.
  Participants
    Female | 188 | 53 | 62 | 303
    Male | 138 | 45 | 34 | 217
Race/Ethnicity, Customized [Number; unit: participants] — The Safety Population (all participants received at least one dose [or any portion of a dose] of study drug) was used for all baseline characteristics.
  participants
    White or Caucasian | 305 | 92 | 93 | 490
    Black or African American | 16 | 5 | 2 | 23
    American Indian or Alaska Native | 1 | 0 | 0 | 1
    Hispanic | 3 | 1 | 1 | 5
    Other, Syrian | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Relapse During the Double-Blind Treatment Period
Description: Relapse was defined as worsening of Restless Legs Syndrome (RLS) symptoms or withdrawal due to lack of efficacy during the 12-week double-blind (DB) treatment period (the period from Randomization on Visit 14 [Week 24] through the end of treatment). Worsening of symptoms was defined as an increase in the total International RLS (IRLS) Scale score by at least 6 or more points relative to the participant's score at Randomization, achieving an IRLS score of at least 15, and an assessment of "much worse" or "very much worse" on the investigator-rated Clinical Global Impression of Change (CGI-C).
Time Frame: DB Treatment Period; Days 169 to 252 (Weeks 24 to 36)
Population: Double-blind Intent-to-Treat (DB ITT) Population: all participants who were randomized into the study, received at least one dose (or any portion of dose) of DB study drug, and for whom at least one post-Randomization visit (Week 24) IRLS Scale total score and investigator-rated CGI-C was available. One participant did not satisfy this description.
Measure: Number; unit: percentage of participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
percentage of participants | 22.7 | 9.4
Statistical Analysis 1: Comparison: DB Placebo vs DB GEn 1200 mg; Test type: Superiority or Other; p = 0.0158, Regression, Logistic — Model included terms for treatment group, randomization IRLS score (Week 24), and pooled study site; Odds Ratio (OR) = 0.353, 95% CI [0.2 to 0.8]

2. Secondary Outcome: Time From Randomization to Relapse in RLS Symptoms During the Double-Blind Treatment Period
Description: Time to relapse was defined as the time until worsening of Restless Legs Syndrome (RLS) symptoms or withdrawal due to lack of efficacy during the 12-week Double-blind (DB) treatment period (same as primary outcome definition). Note: The median is not estimable with Kaplan-Meier methodology when fewer than 50% of participants experience an event. The median is not estimable for this outcome.
Time Frame: DB Treatment Period; Days 169 to 252 (Weeks 24 to 36)
Population: DB ITT Population
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time From Randomization to Relapse in RLS Symptoms During the Double-Blind Treatment Period (Excluding First Two Weeks of DB Phase)
Description: as for outcome 2
Time Frame: DB Treatment Period; Days 184 to 252 (Weeks 26 to 36)
Population: DB ITT Population
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change From Randomization to Week 36 (or End of Treatment) in the IRLS Rating Scale (IRLS) Total Score Using Last Observation Carried Forward (LOCF)
Description: The IRLS Rating scale is a measure of RLS disease severity and reflects the participant-reported assessment of primary sensory and motor features and associated sleep problems in RLS. Items are included that assess the impact of symptoms on participants' mood, daily life, and activities. The total score ranges from 0-40 points, with 40 being the most severe. The scale assesses symptoms over the week prior to measurement. LOCF: Missing data (MD) values were imputed using the last non-missing observation prior to the visit with MD; randomization visit data could be carried forward.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
points on a scale
  Randomization | 5.3 (4.63) | 5.1 (4.20)
  Week 36 | 9.2 (6.76) | 7.0 (7.47)
  Mean change from Randomization to Week 36 | 3.9 (6.49) | 1.9 (7.01)

5. Secondary Outcome: Percentage of Participants Who Responded to Treatment Based on Scores on the Investigator-Rated Clinical Global Impression of Change (CGI-C) Scale as a Dichotomous Variable at Week 36 (DB Treatment Phase) Using LOCF
Description: The CGI-C scale is a widely used tool designed to allow clinicians to rate the severity of illness and the change over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline. For this endpoint, "response" on the CGI-C was defined as participants with a rating of "no change," (score of 4) "minimally improved," (score of 3) "much improved," (score of 2) or "very much improved" (score of 1) compared to Randomization (Week 24).
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
percentage of participants | 67 | 75

6. Secondary Outcome: Number of Participants in Each Category of the Investigator-Rated CGI-C at Week 36 (DB Treatment Phase) Using LOCF
Description: The CGI scale is a widely used tool designed to allow clinicians to rate the severity of illness and the change over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Very much improved (score of 1) | 4 | 10
  Much improved (score of 2) | 5 | 3
  Minimally improved (score of 3) | 12 | 15
  No change (score of 4) | 44 | 44
  Minimally worse (score of 5) | 14 | 13
  Much worse (score of 6) | 11 | 9
  Very much worse (score of 7) | 7 | 2

7. Secondary Outcome: Number of Participants in Each Category of the Participant-Rated CGI-I Scale at Week 36 (DB Treatment Phase) Using LOCF
Description: The participant-rated CGI-I scale is a self-rated assessment designed to allow participants to rate the change of their disease severity over time based on a seven-point scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline.
Time Frame: Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Very much improved (score of 1) | 47 | 60
  Much improved (score of 2) | 30 | 24
  Minimally improved (score of 3) | 7 | 4
  No change (score of 4) | 8 | 6
  Minimally worse (score of 5) | 3 | 0
  Much worse (score of 6) | 1 | 1
  Very much worse (score of 7) | 1 | 1

8. Secondary Outcome: Percentage of Participants Who Responded to Treatment Based on Scores on the Participant-Rated CGI-I at Week 36 (DB Treatment Phase) Using LOCF
Description: The participant-rated CGI-I scale is a self-rated assessment designed to allow participants to rate the change of their disease severity over time based on a seven-point scale, with a score of 1 being "very much improved," and a score of 7 being "very much worse." Response on the participant-rated CGI-I was defined as a rating of "very much improved" (score of 1) or "much improved" (score of 2) compared to Baseline of the SB phase.
Time Frame: Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
percentage of participants | 79.4 | 87.5

9. Secondary Outcome: Mean Change From Randomization to Week 36 (DB Treatment Phase) in the Mean Daytime Somnolence Domain Score of the Medical Outcomes Study (MOS) Sleep Scale Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (hours slept), sleep disturbance, sleep adequacy, and daytime somnolence. Responses are recoded so that a higher score reflects more of the attribute, and then converted to a 0 to 100 scale. The daytime somnolence score is based on questions pertaining to feeling drowsy or sleepy, trouble staying awake, and taking naps > 5 minutes. For daytime somnolence, a negative value indicates an improvement.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
points on a scale
  Randomization | 11.8 (12.20) | 11.0 (14.66)
  Week 36 | 15.5 (16.21) | 12.6 (15.68)
  Change from Randomization to Week 36 | 3.8 (13.33) | 1.5 (11.67)

10. Secondary Outcome: Mean Change From Randomization to Week 36 (DB Treatment Phase) in the Mean Sleep Disturbance Domain Score of the MOS Sleep Scale Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (number of hours slept), sleep disturbance, sleep adequacy, and daytime somnolence. The MOS Sleep Scale sleep disturbance domain is a participant-rated measure of sleep disturbance over the month prior to the measurement. Questions are scored, and responses are converted to a 0 to 100 scale, with lower scores representing less sleep disturbance.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
points on a scale
  Randomization | 16.7 (14.37) | 18.8 (17.21)
  Week 36 | 26.9 (21.24) | 21.0 (19.58)
  Change from Randomization to Week 36 | 10.2 (19.02) | 2.3 (18.32)

11. Secondary Outcome: Change From Randomization to Week 36 (DB Treatment Phase) in the Mean Sleep Adequacy Domain Score of the MOS Sleep Scale Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (number of hours slept), sleep disturbance, sleep adequacy, and daytime somnolence. The MOS Sleep Scale sleep adequacy domain is a participant-rated measure of the adequacy of sleep over the month prior to measurement. Questions are scored, and responses are converted to a 0 to 100 scale, with higher scores representing more adequate ratings of sleep.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
points on a scale
  Randomization | 73.3 (19.30) | 74.6 (21.37)
  Week 36 | 61.6 (28.57) | 70.3 (25.11)
  Change from Randomization to Week 36 | -11.6 (24.01) | -4.3 (22.28)

12. Secondary Outcome: Change From Randomization to Week 36 (DB Treatment Phase) in the Mean Sleep Quantity Domain Score of the MOS Sleep Scale Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (number of hours slept), sleep disturbance, sleep adequacy, and daytime somnolence. The Sleep Quantity Domain score is a participant-rated estimate of the average number of hours of sleep per night over the month.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Groups:
- GEn 1200 mg: Days 169 to 252: two 600 mg ER tablets (1200 mg GEn). Days 253 to 260, participants tapered to one 600 mg ER tablet
Arm/Group | DB Placebo | GEn 1200 mg
Number analyzed (Participants) | 97 | 96
hours
  Randomization | 7.0 (0.95) | 7.0 (0.92)
  Week 36 | 6.8 (1.18) | 6.9 (1.10)
  Change from Randomization to Week 36 | -0.2 (0.90) | -0.1 (0.92)

13. Secondary Outcome: Change From Randomization to Week 36 (DB Treatment Phase) in the RLS Quality of Life (QoL) Overall Life-Impact Score
Description: The RLS QoL is an 18-item scale assessing the impact of RLS on daily life, emotional well-being, social and work life. Responses range from 1 (not at all/never) to 5 (a lot/all of the time). Ten items contribute to a single summary score, the Overall Life Impact, which is standardized to range from 0-100, with lower scores representing better QoL.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
points on a scale
  Randomization | 94.1 (6.74) | 94.3 (6.46)
  Week 36 | 89.9 (12.62) | 92.1 (9.16)
  Change from Randomization to Week 36 | -4.2 (11.53) | -2.2 (7.86)

14. Secondary Outcome: Number of Participants With no Reported RLS Symptoms (Sx) During Each of the 4-hour Periods From the 24-hour RLS Record at Week 36 (DB Treatment Phase)
Description: In the 24-hour RLS Record (diary), participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-minute increments. The period was divided into 7 four-hr intervals (8 AM to 12 PM, 12 to 4 PM, 4 to 8 PM, 6 to 10 PM, 8 to Midnight, Midnight to 4 AM, 4 to 8 AM)
Time Frame: Week 36 (or end of DB treatment)
Population: Double-blind Intent-to-Treat (DB ITT) Population Participants who were missing severity scores for more than two 30-min windows during a 4-hour period had their maximum severity rating for the 4-hour period set to missing. At Randomization (Week 24), there was one participant in each arm with missing 24-hour RLS Record data.
Measure: Number; unit: participants
Groups:
- DB GEn 1200mg: Days 169 to 252: two 600 mg ER tablets (1200 mg GEn). Days 253 to 260, participants tapered to one 600 mg ER tablet
Arm/Group | DB Placebo | DB GEn 1200mg
Number analyzed (Participants) | 96 | 95
participants
  8 AM to 12 PM, Randomization, n=96, 95 | 83 | 88
  8 AM to 12 PM, Week 36, n=87, 89 | 72 | 83
  12 PM to 4 PM, Randomization, n=96, 95 | 85 | 85
  12 PM to 4 PM, Week 36, n=87, 89 | 71 | 78
  4 PM to 8 PM, Randomization, n=96, 95 | 73 | 68
  4 PM to 8 PM, Week 36, n=87, 89 | 68 | 72
  6 PM to 10 PM, Randomization, n=96, 95 | 66 | 61
  6 PM to 10 PM, Week 36, n=87, 89 | 53 | 62
  8 PM to 12 AM, Randomization, n=96, 95 | 62 | 59
  8 PM to 12 AM, Week 36, n=87, 89 | 41 | 61
  12 AM to 4 AM, Randomization, n=96, 95 | 82 | 79
  12 AM to 4 AM, Week 36, n=87, 89 | 66 | 77
  4 AM to 8 AM, Randomization, n=96, 95 | 83 | 83
  4 AM to 8 AM, Week 36, n=87, 89 | 67 | 80

15. Secondary Outcome: Median Time to Onset of First RLS Symptoms Using the 24-hour RLS Symptom Record at Week 36 (DB Treatment Phase)
Description: The 24-hour RLS Record is a diary in which participants report the presence and severity of RLS symptoms (none, mild, moderate, or severe) for a 24-hour period, in 30-min increments beginning at 8AM on the day prior to the visit. Note: The median is not estimable with Kaplan-Meier methodology when fewer than 50% of participants experience an event; thus, no data are presented for the DB GEn 1200 mg arm.
Time Frame: Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 0
hours | 14.5 [13.5 to 17.5] |

16. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire (PSQ) Responses to the Question Regarding Their Overall Quality of Sleep in the Week Prior to Measurement at Randomization and Week 36 (DB Treatment Phase) Using LOCF
Description: The PSQ is designed to evaluate sleep quality, ability to function, and the degree to which RLS symptoms interfere with sleep. Participants rated overall sleep quality and their ability to function on scales ranging from "excellent" to "poor" and were asked to provide the number of nights they experienced RLS symptoms and the number of times/hours they awoke at night during the week prior to the measurement.
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Randomization, Excellent | 38 | 43
  Randomization, Reasonable | 56 | 46
  Randomization, Poor | 3 | 7
  Week 36, Excellent | 29 | 38
  Week 36, Reasonable | 51 | 46
  Week 36, Poor | 17 | 12

17. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire (PSQ) Responses to the Question Regarding Their Ability to Function in the Week Prior to Measurement at Randomization and Week 36 (DB Treatment Phase) Using LOCF
Description: as for outcome 16
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Randomization, Excellent | 53 | 63
  Randomization, Good | 42 | 28
  Randomization, Moderate | 2 | 4
  Randomization, Poor | 0 | 1
  Week 36, Excellent | 44 | 53
  Week 36, Good | 43 | 32
  Week 36, Moderate | 9 | 8
  Week 36, Poor | 1 | 3

18. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Nights With RLS Symptoms in the Week Prior to Measurement at Randomization and Week 36 (DB Treatment Phase) Using LOCF
Description: as for outcome 16
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Randomization, 0 nights | 47 | 38
  Randomization, 1-2 nights | 35 | 36
  Randomization, 3-4 nights | 8 | 11
  Randomization, 5-6 nights | 3 | 5
  Randomization, 7 nights | 4 | 6
  Week 36, 0 nights | 30 | 41
  Week 36, 1-2 nights | 30 | 30
  Week 36, 3-4 nights | 17 | 12
  Week 36, 5-6 nights | 6 | 6
  Week 36, 7 nights | 14 | 7

19. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Awakenings During Night Due to RLS Symptoms in the Week Prior to Measurement at Randomization and Week 36 (DB Treatment Phase) Using LOCF
Description: as for outcome 16
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Randomization, 0 times | 73 | 72
  Randomization, 1-2 times | 22 | 22
  Randomization, 3-4 times | 2 | 1
  Randomization, 5 or more times | 0 | 1
  Week 36, 0 times | 53 | 68
  Week 36, 1-2 times | 35 | 22
  Week 36, 3-4 times | 7 | 5
  Week 36, 5 or more times | 2 | 1

20. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Hours Awake Per Night Due to RLS Symptoms in the Week Prior to Measurement at Randomization and Week 36 (DB Treatment Phase) Using LOCF
Description: as for outcome 16
Time Frame: Randomization (Week 24) and Week 36 (or end of DB treatment)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | DB Placebo | DB GEn 1200 mg
Number analyzed (Participants) | 97 | 96
participants
  Randomization, 0 hours (hr) | 73 | 72
  Randomization, less than 1 hr | 14 | 16
  Randomization, 1 hr to less than 2 hr | 7 | 5
  Randomization, 2 hr to less than 3 hr | 2 | 3
  Randomization, 3 or more hr | 1 | 0
  Week 36, 0 hr | 53 | 68
  Week 36, less than 1 hr | 24 | 17
  Week 36, 1 hr to less than 2 hr | 15 | 8
  Week 36, 2 hr to less than 3 hr | 2 | 3
  Week 36, 3 or more hr | 3 | 0

21. Secondary Outcome: Mean Change From Baseline in the IRLS Scale Total Score at Week 24 (SB Treatment Phase) Using LOCF
Description: The IRLS Rating scale is a measure of disease severity. The scale reflects participant-reported assessment of sensory and motor features and associated sleep problems in RLS. In addition, items are included that assess the impact of symptoms on participants' mood, daily life, and activities. Total score ranges from 0-40 points, with 40 being the most severe.
Time Frame: Days 1 to 168 (Baseline to Week 24 of SB Phase)
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0 through 24) IRLS total score and investigator-rated CGI-I was available. Some participants did not satisfy this description.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
points on a scale
  Baseline | 24.7 (5.48)
  Week 24 | 9.2 (8.35)
  Change from Baseline to Week 24 | -15.5 (9.16)

22. Secondary Outcome: Number of Participants in Each Category of the Investigator-Rated CGI-I at Week 24/End of Treatment (SB Treatment Phase) Using LOCF
Description: The CGI-I scale is a widely used tool designed to allow clinicians to rate the severity of illness and the change over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline.
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Very Much Improved (score of 1) | 170
  Much Improved (score of 2) | 78
  Minimally Improved (score of 3) | 28
  No change (score of 4) | 25
  Minimally worse (score of 5) | 4
  Much Worse (score of 6) | 4
  Very Much Worse (score of 7) | 2

23. Secondary Outcome: Number of Participants in Each Category of the Participant-Rated CGI-I at Week 24/End of Treatment (SB Treatment Phase) Using LOCF
Description: The participant-rated CGI-I scale is a self-rated assessment designed to allow participants to rate the change of their disease severity over time based on a seven-point rating scale, with a score of 1 being "very much improved" and a score of 7 being "very much worse" compared to baseline.
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0-24) IRLS total score and investigator-rated CGI-I was available. Some participants did not satisfy this description and 3 had missing data.
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 308
participants
  Very Much Improved (score of 1) | 163
  Much Improved (score of 2) | 82
  Minimally Improved (score of 3) | 38
  No Change (score of 4) | 16
  Minimally Worse (score of 5) | 7
  Much Worse (score of 6) | 0
  Very Much Worse (score of 7) | 2

24. Secondary Outcome: Mean Change From Baseline to Week 24 (SB Treatment Period) in the Mean Daytime Somnolence Domain Score of the Medical Outcomes Study (MOS) Sleep Scale Using LOCF
Description: as for outcome 9
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0-24) IRLS total score and investigator-rated CGI-I was available. Some participants did not satisfy this description and 12 had missing data.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 299
points on a scale | -21.8 (22.13)

25. Secondary Outcome: Mean Change From Baseline to Week 24 (SB Treatment Period) in the Mean Sleep Disturbance Domain Score of the MOS Sleep Scale Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (number of hours slept), sleep disturbance, sleep adequacy, and daytime somnolence. . The MOS Sleep Scale sleep disturbance domain is a participant-rated measure of sleep disturbance over the month prior to the measurement. Questions are scored, and responses are converted to a 0 to 100 scale, with lower scores representing less sleep disturbance.
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 299
points on a scale | -35.3 (24.92)

26. Secondary Outcome: Mean Change From Baseline to Week 24 (SB Treatment Period) in the Mean Sleep Adequacy Domain Score of the MOS Sleep Scale Using LOCF
Description: as for outcome 11
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 299
points on a scale | 35.7 (30.30)

27. Secondary Outcome: Mean Change From Baseline in the MOS Sleep Scale Domain, Sleep Quantity, Score at Week 24 (SB Treatment Period) Using LOCF
Description: The MOS Sleep Scale is a participant-rated non-disease-specific measure with questions relating to four areas related to sleep: quantity (number of hours slept), sleep disturbance, sleep adequacy, and somnolence. The Sleep Quantity Domain score is a participant-rated estimate of the average number of hours of sleep per night over the month.
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0-24) IRLS total score and investigator-rated CGI-I was available. Some participants did not satisfy this description, and 12 had missing data
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 299
hours | 1.0 (1.45)

28. Secondary Outcome: Mean Change From Baseline in the Overall Quality of Life Impact Score of the RLS Quality of Life (QoL) Questionnaire at Week 24 (SB Treatment Phase)
Description: as for outcome 13
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0-24) IRLS total score and investigator-rated CGI-I was available. Some participants did not satisfy this description, and 13 had missing data
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 298
points on a scale | 25.7 (18.43)

29. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Overall Quality of Sleep in the Week Prior to Measurement at Baseline and Week 24 (SB Treatment Period) Using LOCF
Description: as for outcome 16
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: Single-blind Intent-to-Treat (SB ITT) Population: all participants who enrolled into the study, received at least one dose (or any portion of dose) of SB study drug, and for whom at least one SB visit (Weeks 0-24) IRLS total score and investigator-rated CGI-I was available.
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Baseline, Excellent | 3
  Baseline, Reasonable | 97
  Baseline, Poor | 211
  Week 24, Excellent | 102
  Week 24, Reasonable | 164
  Week 24, Poor | 45

30. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Ability to Function in the Week Prior to Measurement at Baseline and Week 24 (SB Treatment Period) Using LOCF
Description: as for outcome 16
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Baseline, Excellent | 20
  Baseline, Good | 124
  Baseline, Moderate | 141
  Baseline, Poor | 26
  Week 24, Excellent | 145
  Week 24, Good | 127
  Week 24, Moderate | 29
  Week 24, Poor | 10

31. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Nights With RLS Symptoms in the Week Prior to Measurement at Baseline and Week 24 (SB Treatment Period) Using LOCF
Description: as for outcome 16
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Baseline, 0 nights | 1
  Baseline, 1-2 nights | 1
  Baseline 3-4 nights | 36
  Baseline 5-6 nights | 122
  Baseline, 7 nights | 151
  Week 24, 0 nights | 106
  Week 24, 1-2 nights | 98
  Week 24, 3-4 nights | 37
  Week 24, 5-6 nights | 24
  Week 24, 7 nights | 46

32. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Awakenings During the Night Due to RLS Symptoms in the Week Prior to Measurement at Baseline and Week 24 (SB Treatment Period) Using LOCF
Description: as for outcome 16
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Baseline, 0 times | 26
  Baseline, 1-2 times | 131
  Baseline, 3-4 times | 113
  Baseline, 5 or more times | 41
  Week 24, 0 times | 188
  Week 24, 1-2 times | 98
  Week 24, 3-4 times | 18
  Week 24, 5 or more times | 7

33. Secondary Outcome: Number of Participants With the Indicated Post-Sleep Questionnaire Responses to the Question Regarding the Number of Hours Awake Per Night Due to RLS Symptoms in the Week Prior to Measurement at Baseline and Week 24 (SB Treatment Period) Using LOCF
Description: as for outcome 16
Time Frame: Baseline and Day 168 or Week 24/End of Treatment of SB Treatment Phase
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | SB GEn 1200 mg
Number analyzed (Participants) | 311
participants
  Baseline, 0 hours (hr) | 26
  Baseline, less than 1 hr | 78
  Baseline, 1 hr to less than 2 hr | 107
  Baseline, 2 hr to less than 3 hr | 60
  Baseline, 3 or more hr | 40
  Week 24, 0 hr | 188
  Week 24, less than 1 hr | 63
  Week 24, 1 hr to less than 2 hr | 37
  Week 24, 2 hr to less than 3 hr | 17
  Week 24, 3 or more hr | 6

ADVERSE EVENTS:
Time Frame: SB Treatment Emergent Adverse Event (TEAE): Baseline of SB phase through Week 24 including SB taper. DB TEAE: First dose of DB drug (Week 24) through end of DB taper (up to Week 37). SAEs reported up to 30 days after last dose were also reported.
Description: TEAEs were AEs reported in the Safety Population from the time the first dose of study drug was administered in the SB treatment period to the end of the taper period (up to Week 37). AEs were considered TEAEs for the DB treatment period if the onset date or a reported change in severity (for ongoing events) occurred after Randomization.
Arm/Group | SB GEn 1200 mg | DB Placebo | DB GEn 1200 mg
Serious Adverse Events (participants affected / at risk) | 3/326 | 2/98 | 1/96
Other Adverse Events (participants affected / at risk) | 179/326 | 15/98 | 13/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB GEn 1200 mg (N=326) | DB Placebo (N=98) | DB GEn 1200 mg (N=96)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Injury Asphyxiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB GEn 1200 mg (N=326) | DB Placebo (N=98) | DB GEn 1200 mg (N=96)
Somnolence (Nervous system disorders) | 97 (97) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 72 (72) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 41 (41) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 29 (29) | 5 (5) | 3 (3)
Nausea (Gastrointestinal disorders) | 21 (21) | 2 (2) | 3 (3)
Gastroenteritis Viral (Infections and infestations) | 9 (9) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.